CLINICAL TRIAL: NCT04269447
Title: POP-STAR: The Prospective Data Collection on Patients With Abdominal Aortic Aneurysms at the Stockholm Aneurysm Research Group (STAR)
Brief Title: Prospective Aortic Biobank of POP-STAR
Status: Enrolling by invitation | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Rebecka Hultgren, Adjunct Professor, Senior Consultant Vascular Surgery, Karolinska University Hospital
Other Study IDs: EPN201904182
Record Dates: First submitted 2019-12-05; First posted 2020-02-13 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Abdominal Aortic Aneurysm Without Rupture; Abdominal Aortic Aneurysm, Ruptured; Aortic Aneurysm; Aneurysm Abdominal; Aneurysm
Keywords: Growth Prediction; Rupture Risk Prediction; Imaging; Aortic disease; Vascular surgery; Vascular disease; Cardiovascular disease
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Rupture; Aortic Aneurysm; Aneurysm; Aortic Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Structured imaging follow-up — Structured imaging follow-up protocol with ultrasound (US) and computed tomography (CT) examinations as compared to current standard surveillance protocol for individualized estimations of AAA growth.
  Other Names: Finite element analysis (FEA)

SUMMARY:
The overall objective of the POP-STAR project is individualized surveillance for patients diagnosed with abdominal aortic aneurysms by means of more precise, patient-specific AAA growth prediction.

DETAILED DESCRIPTION:
Abdominal aortic aneurysms (AAA, ICD10 I71.4) are asymptomatic dilatations of the infrarenal aorta (≥3cm) with potential to rupture. This multifactorial disease is known to be caused by the progressive degradation of the aortic wall. AAAs have life-threatening consequences in the event of rupture (rAAA): the mortality is 100% if left untreated. The risk of rupture is closely related to the size of the AAA. When a patient is diagnosed with an AAA, life-long surveillance is initiated with regular ultrasound or computed tomography (CT) scans performed at vascular services. Prophylactic surgery is performed when the risk of rupture exceeds the risk of treatment: according to international guidelines, surgical evaluation and repair is indicated at a threshold of 55 mm (50 mm in women) to avoid rupture and subsequent death.

The mortality after planned, elective AAA repair is estimated at 1.5%. By contrast, the mortality after emergency surgery for rAAA reaches 30%. As such, there is much to be gained by early identification of AAAs to enable timely intervention and reduce aneurysm-related morbidity and mortality in the population. The important non-modifiable risk factors for developing the disease include male sex, smoking, high age and family history of AAA. Since 2006, one-time ultrasound screening for AAAs among elderly men has been gradually introduced in Sweden - the programme reached nationwide coverage in 2015. A prevalence of 1.4-2.0% has been recorded in the screened population and an overall reduction of 40% in aneurysm-related death has been demonstrated (annual decline in aneurysm-related mortality of 4%). It is not, however, cost-efficient to screen the female population due to low prevalence and high age at onset of disease.

Previous investigations have indicated that 10-25% of all patients admitted for rupture were already known by the health care system but were subsequently lost to follow-up. Importantly, some large aneurysms never rupture while some small aneurysms (<55 mm) unpredictably do so - in the randomized controlled trial of UKSAT, an annual rupture risk of 1% was documented for small AAAs.

Despite these shortcomings at a patient-specific level, there is still only one verified measure, the diameter, for evaluating growth, risk of rupture and indication for surgery. Consequently, the current follow-up protocol for AAA patients is generalized and fails to consider factors such as age, female sex, smoking, aneurysm morphology and lung function impairment. The major challenge within the field is risk assessment with high precision in order to provide treatment for the right patient and the right time.

The standard surveillance entails repeated diameter measurements: the larger the aneurysm, the shorter the control intervals. The POP-STAR project explores new methods of AAA surveillance by prospective data collection comprising of patient demographics, radiological properties and follow-up information on patients diagnosed with AAAs. All patients will be subjected to standard care flow - POP-STAR adds patient risk profiling and scheduled imaging follow-up. The goal is to be able to characterize the radiological and biomechanical profiles of AAAs for accurate risk stratification, ultimately aiming at individualized AAA patient care.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal aortic aneurysm 35-49 mm in men
* Abdominal aortic aneurysm 30-49 mm in women

Exclusion Criteria:

* Previous aortic or iliac surgery
* Present comorbidities with less than 2-years life expectancy
* Unable or unwilling to give informed consent
* Computed tomography examination with intravenous contrast contraindicated due to renal insufficiency (defined as creatinine/eGFR level XXX)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All men and women diagnosed with an intact abdominal aortic aneurysm (AAA) and who fulfill the inclusion diameter criterion and none of the exclusion criteria are verified at the Department of Vascular Surgery, Karolinska University Hospital, Solna, and consecutively invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Aneurysm expansion rate | Primary outcome evaluated at two years of follow-up.
  Comparison of correctness of predicted growth (diameter vs ASI)
Aneurysm expansion rate | Primary outcome second analysis at two years follow-up.
  Assessment if a more correct predicted growth alters surveillance (ASI vs diameter)

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Department of Vascular Surgery, Karolinska University Hospital, Solna, Stockholm County
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Background] Wanhainen A, Hultgren R, Linne A, Holst J, Gottsater A, Langenskiold M, Smidfelt K, Bjorck M, Svensjo S; Swedish Aneurysm Screening Study Group (SASS). Outcome of the Swedish Nationwide Abdominal Aortic Aneurysm Screening Program. Circulation. 2016 Oct 18;134(16):1141-1148. doi: 10.1161/CIRCULATIONAHA.116.022305. Epub 2016 Sep 14. PMID 27630132
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Sweeting MJ, Thompson SG, Brown LC, Powell JT; RESCAN collaborators. Meta-analysis of individual patient data to examine factors affecting growth and rupture of small abdominal aortic aneurysms. Br J Surg. 2012 May;99(5):655-65. doi: 10.1002/bjs.8707. Epub 2012 Mar 5. PMID 22389113
- [Background] Polzer S, Gasser TC, Vlachovsky R, Kubicek L, Lambert L, Man V, Novak K, Slazansky M, Bursa J, Staffa R. Biomechanical indices are more sensitive than diameter in predicting rupture of asymptomatic abdominal aortic aneurysms. J Vasc Surg. 2020 Feb;71(2):617-626.e6. doi: 10.1016/j.jvs.2019.03.051. Epub 2019 Jun 5. PMID 31176634
- [Background] Polzer S, Gasser TC. Biomechanical rupture risk assessment of abdominal aortic aneurysms based on a novel probabilistic rupture risk index. J R Soc Interface. 2015 Dec 6;12(113):20150852. doi: 10.1098/rsif.2015.0852. PMID 26631334
- [Background] Siika A, Lindquist Liljeqvist M, Zommorodi S, Nilsson O, Andersson P, Gasser TC, Roy J, Hultgren R. A large proportion of patients with small ruptured abdominal aortic aneurysms are women and have chronic obstructive pulmonary disease. PLoS One. 2019 May 28;14(5):e0216558. doi: 10.1371/journal.pone.0216558. eCollection 2019. PMID 31136570
- [Background] Zommorodi S, Roy J, Steuer J, Hultgren R. High proportion of known abdominal aortic aneurysm in patients with rupture indicates surveillance deficiency. J Vasc Surg. 2016 Oct;64(4):949-955.e1. doi: 10.1016/j.jvs.2016.04.007. PMID 27666443
- [Background] Brown LC, Thompson SG, Greenhalgh RM, Powell JT; UK Small Aneurysm Trial Participants. Fit patients with small abdominal aortic aneurysms (AAAs) do not benefit from early intervention. J Vasc Surg. 2008 Dec;48(6):1375-81. doi: 10.1016/j.jvs.2008.07.014. PMID 19118733
- [Background] Singh K, Bonaa KH, Jacobsen BK, Bjork L, Solberg S. Prevalence of and risk factors for abdominal aortic aneurysms in a population-based study : The Tromso Study. Am J Epidemiol. 2001 Aug 1;154(3):236-44. doi: 10.1093/aje/154.3.236. PMID 11479188
- [Background] Scott RA, Bridgewater SG, Ashton HA. Randomized clinical trial of screening for abdominal aortic aneurysm in women. Br J Surg. 2002 Mar;89(3):283-5. doi: 10.1046/j.0007-1323.2001.02014.x. PMID 11872050
- [Background] Sakalihasan N, Michel JB, Katsargyris A, Kuivaniemi H, Defraigne JO, Nchimi A, Powell JT, Yoshimura K, Hultgren R. Abdominal aortic aneurysms. Nat Rev Dis Primers. 2018 Oct 18;4(1):34. doi: 10.1038/s41572-018-0030-7. PMID 30337540